CLINICAL TRIAL: NCT00498875
Title: Depression and Adherence in Head and Neck Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2004-0390; NCI-2012-02098 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-06; First posted 2007-07-10 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Oropharyngeal Cancer; Head and Neck Cancer
Keywords: Oropharyngeal Cancer; Head and Neck Cancer; Depression; Questionnaire; Survey; Interview
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire + Depression Intervention
  Interventions: Behavioral: Questionnaire; Behavioral: Depression Intervention

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire regarding mood, coping with cancer, how closely you follow your treatment schedule, your thoughts, your demographic information (such as age and race), and your medical history. If the answers to your questionnaire indicate that you may be depressed, you will be offered the intervention portion of the study.
  Other Names: Survey
Behavioral: Depression Intervention — Sessions given over 7 weeks and each lasting 30-45 minutes, that use "cognitive-behavioral" techniques.

SUMMARY:
Primary Objectives:

* Develop and pilot test an innovative intervention to determine its feasibility and acceptability to patients. Recruitment rate, patient satisfaction, attendance, questionnaire completion rates and the reliability and validity of the questionnaires will be assessed.
* Conduct preliminary analyses on the efficacy of the intervention in improving patients' depression. Evaluate whether depression levels in patients receiving the intervention decreases, and whether the decrease is greater among those who complete more sessions.
* Test the relationship between patients' depression levels and adherence to swallowing rehabilitation and to dental preventive maintenance regimens.

DETAILED DESCRIPTION:
You will be asked to fill out a questionnaire containing questions about your mood, coping with cancer, how closely you follow your treatment schedule, your thoughts, your demographic information (such as age and race), and your medical history. It should take between 25-35 minutes to complete the questionnaire. If you score as nondepressed on the questionnaire, you will be contacted again every week for 6 weeks during radiation treatment, to check for depression again. If you score as depressed during a later screening, you will then be asked additional questions about your symptoms, coping, and social support. It should take between 10-20 minutes to complete these additional questions.

If the answers to your questionnaire indicate that you may be depressed, you will be offered the intervention portion of the study. Only those participants who score as depressed on the questionnaire will be assigned to the intervention. You will then be informed of your test results, and provided with a list of community referrals. Whoever is responsible for your treatment, whether he or she is a M.D. Anderson physician, community referring physician, or both, will also be informed of these test results, and a note will be added to your medical record.

You will be asked to take part in 7 sessions with a trained doctoral-level psychologist or advanced clinical doctoral student under the supervision of a licensed psychiatrist. The first two sessions may be conducted in person, face to face, or may be conducted over the telephone. The remaining five sessions will be done over the telephone. These sessions will last between 30 and 45 minutes and will occur every week for seven weeks.

The 30-45 minute telephone sessions will use "cognitive-behavioral" techniques, a method proven to be effective in relieving depressive symptoms. Cognitive-behavioral techniques will teach you skills in relaxation and activity scheduling, as well as ways to recognize and fight negative thoughts. You will also be given a journal to record and practice ways of fighting depression. The intervention will include an educational component for your spouse/partner or caregiver on the nature of clinical depression. The spouse/caregiver will be given a booklet which explains facts about depressive disorders and helpful ways that they can support you. You may also be given over-the counter samples of toothpaste and oral products if approved by your doctor or dentist. You will also be given the use of a mini-food-blender to help you problem solve issues of eating during the course of the study. You will be asked to return the mini-food-blender at the end of the study.

If you participate in the intervention, upon completion, you will receive a short survey asking about your satisfaction with the intervention. After completing the first questionnaire, you may be contacted again to complete five follow-up questionnaires, at the beginning of radiation treatment, as well as, six and twelve weeks and again, six and twelve months after radiation treatment begins. The questionnaires will be similar to the first one but will also contain questions about any additional depression care you received while participating in the study or after the intervention. This information will include prescription of antidepressants, formal referral to psychiatric services, referral to support groups, and any depression care you received in addition to the intervention in this study. You will also be asked how closely you followed the swallowing exercises, your dental care habits, and your referrals to other sources in the community.

Researchers will also collect medical information from your medical record such as cancer stage, if the disease has gotten worse, treatment, and side effects. This information will allow researchers to look at how specific treatments affect patients. You may also be involved in an interview regarding your personal experience. The study staff will tape-record the interview after you have given your consent verbally and on the tape. In order to protect your confidentiality, the study staff will store the digital record of the interview on an external hard drive, and the record will be destroyed after the study is complete.

To provide quality control for the intervention, a random sample of telephone counseling sessions may be tape-recorded. Before tape-recording the session, the counselor will ask for your permission to be tape-recorded, and will then tape-record your permission on the audiotape. No identifying information will be recorded on the audiotape, and the recorded sessions will be reviewed by project team members for research purposes only. Audiotapes will be labeled with study identification numbers only, so none of your personal information will be on the tape itself.

If your answers to the questionnaires or your responses during the face-to-face sessions or telephone calls show that you are having suicidal thoughts or may need antidepressant medication, you will be referred for a consultation with Dr. Alan Valentine, a M.D. Anderson psychiatrist who is also participating in this research study. Researchers will also let your treating physicians know about the referral to Dr. Valentine, if you are referred for further treatment.

If your answers to the questionnaires or your responses during the face to face sessions or telephone calls show that you have a problem with alcohol abuse, you will be referred for a consultation with Dr. Kathleen Rickman, a M.D. Anderson advanced nurse practitioner who is also participating in this research study. Researchers will also let your treating physicians know about the referral to Dr. Rickman if you are referred for further treatment.

This is an investigational study. A total of 350 head and neck cancer patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I-IV
2. At least 18 years of age
3. Speak and read English at a 7th grade level
4. Are oriented to time, person, and place
5. Have a Zubrod performance status of 0-3.
6. To be eligible for the pilot depression intervention patients must score 9 or above on the Patient Health Questionnaire (PHQ-9). Additionally, if a patient has an elevated PHQ score and does not meet the cutoff but expresses a desire to be in the intervention in order to relieve his or her depression, then the PI will contact the participant to further assess eligibility for the intervention. Patients who do not make the cut-off will still be included in the study's statistical analyses.

Exclusion Criteria:

1. Do not have other cancer diagnoses, excepting non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants with stage I-IV Head and Neck Cancer.
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2005-03-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate, Patient satisfaction, Attendance, Questionnaire Completion Rates (questionnaire responses) | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Eileen H. Shinn, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org